CLINICAL TRIAL: NCT04699812
Title: Atrial Fibrillation Algorithms Clinical Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apple Inc. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 099-25141
Record Dates: First submitted 2020-12-04; First posted 2021-01-07 (Actual); Results first posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
Keywords: CARDIOVASCULAR DISEASES; HEART DISEASES; ARRHYTHMIA; CARDIAC
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases; Arrhythmias, Cardiac | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- COHORT 1 (Other): This will include subjects with no known history of AF
  Interventions: Device: ELECTROCARDIOGRAM (ECG) PATCH WEAR
- COHORT 2 (Other): This will include subjects with no known history of aF, but with history of frequent premature atrial contractions (PACs), frequent premature ventricular contractions (PVCs), supraventricular tachycardia (SVT), or non-sustained ventricular tachycardia (NSVT)
  Interventions: Device: ELECTROCARDIOGRAM (ECG) PATCH WEAR
- COHORT 3 (Other): This will include subjects with known history of paroxysmal, persistent, or chronic AF
  Interventions: Device: ELECTROCARDIOGRAM (ECG) PATCH WEAR
- COHORT 4 (Other): Will include subjects with permanent AF
  Interventions: Device: ELECTROCARDIOGRAM (ECG) PATCH WEAR

INTERVENTIONS:
Device: ELECTROCARDIOGRAM (ECG) PATCH WEAR — ALL PARTICIPANTS WILL WEAR AN ECG PATCH ON THEIR UPPER LEFT CHEST THROUGHOUT THE STUDY PARTICIPATION
  Other Names: CARDEASOLO

SUMMARY:
The purpose of the study is to evaluate the performances of investigational Irregular Rhythm Notification Feature (version 2.0) and Atrial Fibrillation History Feature algorithms.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the performances of investigational Irregular Rhythm Notification Feature (version 2.0) and Atrial Fibrillation History Feature algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and provide written informed consent
2. Willing and able to participate in the study procedures as described in the consent form
3. Be 22 years of age and older
4. Able to communicate effectively with and follow instructions from the study staff
5. Able to wear the wrist device for duration of study participation
6. For Cohort 1, have no known medical history of AF
7. For Cohort 2, have no known medical history of AF and active diagnosis of at least one of the following arrhythmias within the past 2 years:

   1. Frequent PACs, defined as at least 1% of total beats of atrial ectopic beats by 24-48 hour Holter, ambulatory ECG monitor, or implantable loop recorder)
   2. Frequent PVCs, defined as at least 1% of total beats of ventricular ectopic beats by 24-48 hour Holter, ambulatory ECG monitor, or implantable loop recorder
   3. SVT, which will include atrial tachycardia, atrioventricular nodal re-entrant tachycardia, atrioventricular re-entrant tachycardia by 12-lead ECG or 24-48 hour Holter, ambulatory ECG monitor, or implantable loop recorder
   4. NSVT, defined as three or more consecutive ventricular beats at a rate of at least 100 beats per minute and lasting no more than 30 seconds, by 12-lead ECG or 24-48 hour Holter, ambulatory ECG monitor, or implantable loop recorder
8. For Cohorts 3 and 4, have a known diagnosis of AF at the time of screening (confirmed by electronic medical record (EMR) or self-report) and have had a recent episode of AF, or confirmed AF on ECG, in the past 12 months
9. For Cohort 4, have a known diagnosis of permanent AF at the time of screening (confirmed by EMR or self-report) and have had a recent episode of AF, or confirmed AF on ECG, in the past 12 months
10. Meet additional binning based on demographics.

Exclusion Criteria:

1. Physical disability that precludes safe and adequate testing
2. Mental impairment resulting in limited ability to cooperate
3. Known uncontrolled medical conditions, such as (but not limited to) significant anemia, important electrolyte imbalance and untreated or uncontrolled thyroid disease
4. Open wound(s) on the wrist and/or forearm
5. Tattoos, large moles, or scars on the wrist at the wrist device location
6. Skin conditions on either wrist that would preclude subject from wearing a wristband on either wrist
7. Known allergy or sensitivity to medical adhesives, isopropyl alcohol, wristbands, or ECG patch
8. Medical history or physical assessment finding that makes the subject inappropriate for participation according to investigator(s)
9. Participation in a previous study that used a wrist-worn sensor device with a simultaneous ECG reference patch
10. Implantable cardiac devices such as a Pacemaker or Implantable Cardioverter Defibrillator
11. Clinically significant hand tremors, as judged by the investigator
12. Acute illness including COVID and other respiratory illnesses
13. Subjects with known history of AF on rhythm control medications with history of complete AF rhythm control (i.e history of zero AF burden) will be excluded from Cohorts 3 and 4

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Tsay, MD, PhD, Study Director — Apple Inc.
Locations (4):
- United States (4):
  - Clinical Research of South Florida, Coral Gables, Florida
  - American Health Network of Indiana Llc, Avon, Indiana
  - Heartland Cardiology Webb, Wichita, Kansas
  - Healtheast, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4
Started | 78 | 82 | 366 | 47
Completed | 70 | 64 | 304 | 45
Not Completed | 8 | 18 | 62 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Total
Number analyzed (Participants) | 78 | 82 | 366 | 47 | 573
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 45 | 144 | 14 | 263
  >=65 years | 18 | 37 | 222 | 33 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (16.68) | 61.2 (15.07) | 65.4 (11.79) | 70.0 (8.85) | 63.0 (14.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 53 | 180 | 14 | 287
  Male | 38 | 29 | 186 | 33 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 1 | 17 | 2 | 38
  Not Hispanic or Latino | 60 | 81 | 349 | 45 | 535
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 1 | 5
  Asian | 0 | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 7 | 27 | 4 | 57
  White | 57 | 74 | 330 | 41 | 502
  More than one race | 0 | 0 | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78 | 82 | 366 | 47 | 573

OUTCOME MEASURES:

1. Primary Outcome: SENSITIVITY OF IRREGULAR RHYTHM NOTIFICATION FEATURE [IRNF]
Description: Sensitivity of the irregular rhythm notification for the identification of persons with AF by 13-day ambulatory ECG, with AF defined as at least 30 seconds of AF by ambulatory ECG. Sensitivity is defined as the percentage of subjects exhibiting AF on the ambulatory ECG who also received an irregular rhythm notification concordant with at least one episode of AF.
Time Frame: 13 DAYS
Population: Per the pre-specified analysis plan, subjects from only Cohorts 1, 3, and 4 were to be included in the analysis. The pre-specified analysis also required the results to be pooled across these 3 cohorts and were not to be reported separately by cohort.
Measure: Number; unit: percentage of participants
Groups:
- Overall: Pooled across relevant cohorts per the statistical analysis section of the protocol.
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 1 | 0 | 103 | 36 | 140
percentage of participants | NA — Cohort not analyzed separately per statistical analysis section of the protocol. |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 88.6

2. Primary Outcome: SPECIFICITY OF LACK OF IRREGULAR RHYTHM NOTIFICATIONS FEATURE [IRNF]
Description: Specificity of the lack of irregular rhythm notification for the identification of persons without AF by 13-day ambulatory ECG, with AF defined as at least 30 seconds of AF by ambulatory ECG. Specificity is defined as the percentage of subjects not exhibiting AF on the ambulatory ECG who also did not receive any irregular rhythm notifications.
Time Frame: 13 DAYS
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 66 | 0 | 219 | 7 | 292
percentage of participants | NA — Cohort not analyzed separately per statistical analysis section of the protocol. |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 99.3

3. Primary Outcome: WEEKLY ATRIAL FIBRILLATION BURDEN FEATURE ESTIMATE [AFBF]
Description: Weekly AF burden estimate defined as the percentage of time a subject is in Atrial Fibrillation during wrist device wear over the prior 7 consecutive days. The weekly AF burden was estimated by both the reference device and the algorithm and reported using the Bland-Altman limits of Agreement.
Time Frame: 13 DAYS
Population: Per the pre-specified analysis plan, subjects from only Cohorts 3 and 4 (i.e., those with a prior diagnosis of AF) were to be included in the analysis. The pre-specified analysis also required the results to be pooled across these 2 cohorts and were not to be reported separately by cohort.
Measure: Number; unit: Bland-Altman Limits of Agreement
Units Other Than Participants: Paired Differences
Arm/Group | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 244 | 36 | 280
Number analyzed (Paired Differences) | 244 | 36 | 280
Bland-Altman Limits of Agreement
  Lower Limit of Agreement (%) | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | -11.4
  Upper Limit of Agreement (%) | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 12.8

4. Secondary Outcome: POSITIVE PREDICTIVE VALUE OF IRREGULAR RHYTHM NOTIFICATION FEATURE [IRNF]
Description: Notification-level positive predictive value (PPV) with AF by ambulatory ECG at the time of any tachogram comprising the notification.
Time Frame: 13 DAYS
Population: Per the pre-specified analysis plan, subjects from only Cohorts 1, 3 and 4 who received a notification were to be included in the analysis. No subjects in Cohort 1 received a notification in the study. The pre-specified analysis also required the results to be pooled across the cohorts and were not to be reported separately by cohort.
Measure: Number; unit: percentage of notifications
Units Other Than Participants: Notifications
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 0 | 0 | 92 | 35 | 127
Number analyzed (Notifications) | 0 | 0 | 1228 | 617 | 1845
percentage of notifications |  |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 100

5. Secondary Outcome: TACHOGRAM ALERT SENSITIVITY [IRNF]
Description: Tachogram-level sensitivity performance for tachograms comprising alerts.
Time Frame: 13 DAYS
Population: Per the pre-specified analysis plan, subjects from only Cohorts 1, 3 and 4 were to be included in the analysis if they received a notification during the study. No subjects in Cohort 1 received a notification. The pre-specified analysis also required the results to be pooled across the cohorts and were not to be reported separately by cohort.
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 0 | 0 | 92 | 35 | 127
Number analyzed (Tachograms) | 0 | 0 | 7013 | 3518 | 10531
percentage of tachograms |  |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 95.05

6. Secondary Outcome: TACHOGRAM ALERT SPECIFICITY [IRNF]
Description: Tachogram-level specificity performance for tachograms comprising alerts.
Time Frame: 13 DAYS
Population: Per the pre-specified analysis plan, subjects from only Cohorts 1, 3 and 4 were to be included in the analysis if they received a notification. No subjects in Cohort 1 received a notification during the study. The pre-specified analysis also required the results to be pooled across the cohorts and were not to be reported separately by cohort.
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 5
Number analyzed (Tachograms) | 0 | 0 | 2 | 5 | 7
percentage of tachograms |  |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 0

7. Secondary Outcome: Tachogram Alert False Positive Rate [IRNF]
Description: Tachogram-level False Positive rate performance for tachograms comprising alerts.
Time Frame: 13 DAYS
Population: as for outcome 6
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 0 | 0 | 8 | 6 | 14
Number analyzed (Tachograms) | 0 | 0 | 8 | 9 | 17
percentage of tachograms |  |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 100

8. Secondary Outcome: Tachogram Alert Positive Predictive Value [IRNF]
Description: Tachogram-level Positive Predictive value performance for tachograms comprising alerts.
Time Frame: 13 DAYS
Population: as for outcome 6
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 0 | 0 | 92 | 35 | 127
Number analyzed (Tachograms) | 0 | 0 | 6672 | 3355 | 10027
percentage of tachograms |  |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 99.83

9. Secondary Outcome: Tachogram Alert Negative Predictive Value [IRNF]
Description: Tachogram-level Negative Predictive value performance for tachograms comprising alerts.
Time Frame: 13 DAYS
Population: as for outcome 6
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 0 | 0 | 78 | 33 | 111
Number analyzed (Tachograms) | 0 | 0 | 349 | 172 | 521
percentage of tachograms |  |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 0

10. Secondary Outcome: TACHOGRAM SENSITIVITY [IRNF]
Description: Tachogram-level sensitivity performance for all generated tachograms.
Time Frame: 13 DAYS
Population: Per the pre-specified analysis plan, subjects from only Cohorts 1, 3 and 4 were to be included in the analysis. The pre-specified analysis also required the results to be pooled across the cohorts and were not to be reported separately by cohort.
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 8 | 0 | 131 | 38 | 177
Number analyzed (Tachograms) | 8 | 0 | 2818 | 1663 | 4489
percentage of tachograms | NA — Cohort not analyzed separately per statistical analysis section of the protocol. |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 85.5

11. Secondary Outcome: TACHOGRAM SPECIFICITY [IRNF]
Description: Tachogram-level specificity performance for all generated tachograms.
Time Frame: 13 DAYS
Population: as for outcome 10
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 68 | 0 | 265 | 10 | 343
Number analyzed (Tachograms) | 685 | 0 | 2578 | 90 | 3353
percentage of tachograms | NA — Cohort not analyzed separately per statistical analysis section of the protocol. |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 99.9

12. Secondary Outcome: TACHOGRAM FALSE POSITIVE RATE [IRNF]
Description: Tachogram-level false positive rate performance for all generated tachograms.
Time Frame: 13 DAYS
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Groups:
- Overall: Pooled across relevant cohorts per statistical analysis section of the protocol.
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 68 | 72 | 269 | 12 | 349
Number analyzed (Tachograms) | 726 | 5937 | 2823 | 104 | 3653
percentage of tachograms | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 0.05 | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 0.22

13. Secondary Outcome: TACHOGRAM POSITIVE PREDICTIVE VALUE [IRNF]
Description: Tachogram-level positive predictive value performance for all generated tachograms.
Time Frame: 13 DAYS
Population: Per the pre-specified analysis plan, subjects from only Cohorts 1, 3 and 4 were to be included in the analysis if they had at least one irregular tachogram. No subjects in Cohort 1 had an irregular tachogram. The pre-specified analysis also required the results to be pooled across the cohorts and were not to be reported separately by cohort.
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 0 | 0 | 93 | 36 | 129
Number analyzed (Tachograms) | 0 | 0 | 2370 | 1474 | 3844
percentage of tachograms |  |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 99.8

14. Secondary Outcome: TACHOGRAM NEGATIVE PREDICTIVE VALUE [IRNF]
Description: Tachogram-level negative predictive value performance for all generated tachograms.
Time Frame: 13 DAYS
Population: as for outcome 10
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 68 | 0 | 322 | 43 | 433
Number analyzed (Tachograms) | 734 | 0 | 3271 | 293 | 4298
percentage of tachograms | NA — Cohort not analyzed separately per statistical analysis section of the protocol. |  | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 77.9

15. Secondary Outcome: TACHOGRAM SENSITIVITY [AFBF]
Description: Sensitivity of tachograms for the identification of AF by ambulatory ECG.
Time Frame: 13 days
Population: Per the pre-specified analysis plan, subjects from only Cohorts 3 and 4 (i.e., those with a prior diagnosis of AF) were to be included in the analysis. The pre-specified analysis also required the results to be pooled across the cohorts and were not to be reported separately by cohort.
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 135 | 42 | 177
Number analyzed (Tachograms) | 1412 | 758 | 2170
percentage of tachograms | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 92.6

16. Secondary Outcome: TACHOGRAM SPECIFICITY [AFBF]
Description: Specificity of tachograms for the identification of AF by ambulatory ECG.
Time Frame: 13 days
Population: as for outcome 15
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 273 | 13 | 286
Number analyzed (Tachograms) | 5333 | 125 | 5458
percentage of tachograms | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 98.8

17. Secondary Outcome: TACHOGRAM POSITIVE PREDICTIVE VALUE [AFBF]
Description: Positive Predictive Value of tachograms for the identification of AF by ambulatory ECG.
Time Frame: 13 days
Population: as for outcome 15
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 111 | 40 | 151
Number analyzed (Tachograms) | 1331 | 746 | 2077
percentage of tachograms | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 96.7

18. Secondary Outcome: TACHOGRAM NEGATIVE PREDICTIVE VALUE [AFBF]
Description: Negative Predictive Value of tachograms for the identification of AF by ambulatory ECG.
Time Frame: 13 days
Population: as for outcome 15
Measure: Number; unit: percentage of tachograms
Units Other Than Participants: Tachograms
Arm/Group | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 272 | 11 | 283
Number analyzed (Tachograms) | 5414 | 137 | 5551
percentage of tachograms | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 97.1

19. Secondary Outcome: DAY-SPECIFIC AF BURDEN ESTIMATE [AFBF]
Description: Day-specific AF burden estimate defined as the percentage of time a subject is in Atrial Fibrillation during a specific day of the week.
Time Frame: 13 DAYS
Population: as for outcome 15
Measure: Number; unit: percent of iterations achieving success
Units Other Than Participants: Simulation Iterations
Arm/Group | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 256 | 34 | 290
Number analyzed (Simulation Iterations) | 2000 | 2000 | 2000
percent of iterations achieving success | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 62.5

20. Secondary Outcome: FOUR-HOUR SEGMENT SPECIFIC AF BURDEN ESTIMATE [AFBF]
Description: Four-hour segment-specific AF burden estimate defined as the percentage of time a subject is in Atrial Fibrillation during a specific four-hour segment of a day
Time Frame: 13 DAYS
Population: as for outcome 15
Measure: Number; unit: percent of iterations achieving success
Units Other Than Participants: Simulation Iterations
Arm/Group | COHORT 3 | COHORT 4 | Overall
Number analyzed (Participants) | 291 | 38 | 329
Number analyzed (Simulation Iterations) | 2000 | 2000 | 2000
percent of iterations achieving success | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | NA — Cohort not analyzed separately per statistical analysis section of the protocol. | 99.95

ADVERSE EVENTS:
Time Frame: 3.5 months
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/82 | 0/366 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/82 | 7/366 | 0/47
Other Adverse Events (participants affected / at risk) | 3/78 | 11/82 | 46/366 | 3/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1 (N=78) | COHORT 2 (N=82) | COHORT 3 (N=366) | COHORT 4 (N=47)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 (1) | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 (1) | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Dementia/Asthenia (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1 (N=78) | COHORT 2 (N=82) | COHORT 3 (N=366) | COHORT 4 (N=47)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 3 (3) | 11 (11) | 46 (46) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT04699812/Prot_SAP_000.pdf